CLINICAL TRIAL: NCT03412591
Title: The Efficacy of Suvorexant in the Residential Treatment of Patients With Substance Use Disorder and Insomnia: A Pilot Open Trial
Brief Title: The Efficacy of Suvorexant in Treatment of Patients With Substance Use Disorder and Insomnia: A Pilot Open Trial
Acronym: Suvsubuse
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Scott C Bunce, PhD, Associate Professor of Psychiatry, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00005409
Record Dates: First submitted 2017-11-27; First posted 2018-01-26 (Actual); Results first posted 2024-02-12 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Sleep Disturbance; Craving; Cortisol; Hypersecretion
MeSH Terms: conditions — Parasomnias | interventions — suvorexant

STUDY DESIGN:
Intervention Model Description: We intend to evaluate the efficacy of suvorexant in a group of opioid dependent (n=14) and a group of alcohol dependent subjects (n=14) in a residential treatment facility. It is an open label trial on subjects with opioid or alcohol dependence who are 5to 10 days post withdrawal.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Open label trial of suvorexant in individuals with opioid use disorder (Other): It is an open label trial to study the efficacy of suvorexant in a group of patients with opioid use disorder.
  Interventions: Drug: Suvorexant 20 mg
- Open label trial of suvorexant in individuals with alcohol use disorder (Other): It is an open label trial to study the efficacy of suvorexant in a group of patients with alcohol use disorder.
  Interventions: Drug: Suvorexant 20 mg

INTERVENTIONS:
Drug: Suvorexant 20 mg — Suvorexant 20 mg is an orexin 1/2receptor antagonist approved for the treatment of sleep disturbance in subjects with Primary Insomnia.
  Other Names: Belsomra

SUMMARY:
Insomnia is an extremely common and poorly treated problem in patients with substance use disorders (SUD)s undergoing rehabilitation treatment in a residential facility. The persistence of insomnia in substance use disorders (SUDs) may be associated with tonic levels of drug craving. Insomnia and craving can predispose to relapse in patients with SUDs. Insomnia and SUDs are independently associated with increased cortisol indicating physiological dysregulation of the stress response system including the hypothalamic-pituitary-adrenal (HPA) axis. Hence sleep disturbance, craving and increased cortisol leads to relapse in SUD subjects. Suvorexant, an orexin 1 / 2 receptor antagonist, approved by the FDA for the treatment of sleep disturbance in subjects with primary Insomnia. Previous animal studies report Orexin 1 receptor antagonist decreases craving and normal the HPA axis. However, the efficacy of suvorexant on sleep and craving in SUD subjects is not known. The primary aims of this study are-

1. To determine if suvorexant will improve sleep quality (increased total sleep time, fewer awakenings), as measured through wrist actigraphy and the Insomnia Severity Index (ISI) in SUDs.
2. To assess whether or not SUDs patients treated with suvorexant endorse scale items on a modified abuse liability assessment battery.
3. To determine if daily reports of mood, stress, craving and sleep using Ecological Momentary Assessment (EMA data) change during the course of the study as patients with SUDs are treated with suvorexant.
4. To determine if patients taking suvorexant will have a decrease in total daily salivary cortisol over the course of the study by collecting samples at five time points in a day, for two consecutive days at two different times in the study.

DETAILED DESCRIPTION:
Insomnia is an extremely common and poorly treated problem in patients with substance use disorders (SUD)s patients undergoing rehabilitation treatment in residential facility. The persistence of insomnia in substance use disorders (SUDs) may be associated with tonic levels of drug craving. Insomnia and craving can predispose to relapse in patients with SUDs. Insomnia and SUDs are independently associated with increased cortisol indicating physiological dysregulation of the stress response system including the hypothalamic-pituitary-adrenal (HPA) axis. Hence sleep disturbance, craving and increased cortisol leads to relapse in SUD subjects.

Suvorexant is a novel orexin 1 and 2 receptor antagonist, FDA approved for the treatment of insomnia. Suvorexant may be differentially beneficial in patients with opioid dependence: 1) It is efficacious for treatment of insomnia in the general population, 2) Data from animal models of opioid dependence suggest that orexins may be involved in reward (opioid) seeking behavior and altered stress response while an orexin antagonist appears to decrease reward (opioid) seeking while normalizing HPA axis function. A medication that can improve sleep, decrease craving and normalize the HPA axis may theoretically be helpful in patients with SUDs. At this juncture, the literature supports the case for an open trial of Suvorexant for patients in residential care for SUDs, who complain of sleep disturbance. The patients will be at least 5 days post-withdrawal, in order to minimize the residual sleep complaints associated with that phase of treatment.

In previous, well-designed, placebo-controlled clinical trials in patients with insomnia, suvorexant has been shown to be efficacious compared with placebo. However, substance dependent patients with insomnia were not included in these studies. Although, as a new sleep medication, suvorexant has been placed in Schedule IV by the FDA, the drug has not been studied in the context of its potential abuse liability when administered at bedtime at the therapeutic dose among patients in residential treatment for substance dependence disorders. A modified abuse liability protocol will therefore be incorporated in this pilot study.

The hypothesis for this study are-

1. Relative to a baseline, patients treated with suvorexant will experience an increase in total sleep time, fewer awakenings after sleep onset, and improved subjective sleep quality.
2. Patients treated with suvorexant are not likely to endorse scale items associated with abuse liability 30 minutes after drug administration or the following morning.
3. Relative to baseline, patients being treated with suvorexant are more likely to report improved moods, and decreased ambient craving.
4. Relative to baseline, patients being treated with suvorexant are more likely to experience decreased total daily salivary cortisol over the course of 7 days of treatment with suvorexant.

ELIGIBILITY:
Inclusion Criteria:

1. Sex: male or female
2. Age: 21-64 (inclusive) years old
3. Caron Foundation residential alcohol or opioid dependent patients that have a history of daily or near daily substance use for the month prior to admittance.

   Group 1: at least five days post medically assisted withdrawal for alcohol dependence, and complain of problems falling asleep, remaining asleep after sleep onset, or poor sleep quality on current sleep medication (antidepressant/melatonin).

   Group 2: at least five days post medically assisted withdrawal for opioid dependence and complain of problems falling asleep, remaining asleep after sleep onset, or poor sleep quality on current sleep medication (antidepressant/melatonin).
4. Fluent in written and spoken English.

Exclusion Criteria:

1. Patients who are concurrently receiving a psychoactive drug for the treatment of an Axis I disorder excluding sedating antidepressants that have been prescribed for the treatment of sleep disturbance.
2. Patients with current major depressive disorder, schizophrenia, bipolar disorder, post traumatic stress disorder, or a history of traumatic brain injury.
3. Patients with a history of narcolepsy or REM related phenomenon.
4. Patients with chronic respiratory problems including asthma, COPD, or other respiratory issues that can lead to sleep disturbances at night.
5. Patients with current suicidal ideation, or a history of previous suicide attempts.
6. Patients with severe liver impairment.
7. Women who are pregnant or breastfeeding.
8. Patients who are severely obese.
9. Decisional impairment
10. Prisoners or under legal mandate.

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2023-01-07 (Actual); Study Completion 2023-01-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Venkatesh Basappa Krishnamurthy, MD, Principal Investigator — Penn State University Hershey Medical Center
Locations (1):
- Richard J Caron Foundation, Wernersville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] US Food and Drug Administration (2013). Suvorexant Advisory Committee Meeting briefing document.http://www.fda.gov/downloads/advisorycommittees/committeesmeetingmaterials/drugs/peripheralandcentralnervoussystemdrugsadvisorycommittee/ucm352970.pdf. Accessed 9 Sep 2014
- [Background] Smith RJ, Aston-Jones G. Orexin / hypocretin 1 receptor antagonist reduces heroin self-administration and cue-induced heroin seeking. Eur J Neurosci. 2012 Mar;35(5):798-804. doi: 10.1111/j.1460-9568.2012.08013.x. Epub 2012 Feb 22. PMID 22356621
- [Background] Giardino WJ, de Lecea L. Hypocretin (orexin) neuromodulation of stress and reward pathways. Curr Opin Neurobiol. 2014 Dec;29:103-8. doi: 10.1016/j.conb.2014.07.006. Epub 2014 Jul 20. PMID 25050887
- [Background] Koob G, Kreek MJ. Stress, dysregulation of drug reward pathways, and the transition to drug dependence. Am J Psychiatry. 2007 Aug;164(8):1149-59. doi: 10.1176/appi.ajp.2007.05030503. PMID 17671276
- [Background] Goldstein RZ, Volkow ND. Dysfunction of the prefrontal cortex in addiction: neuroimaging findings and clinical implications. Nat Rev Neurosci. 2011 Oct 20;12(11):652-69. doi: 10.1038/nrn3119. PMID 22011681
- [Background] Brower KJ. Alcohol's effects on sleep in alcoholics. Alcohol Res Health. 2001;25(2):110-25. PMID 11584550
- [Background] Conroy DA, Arnedt JT. Sleep and substance use disorders: an update. Curr Psychiatry Rep. 2014 Oct;16(10):487. doi: 10.1007/s11920-014-0487-3. PMID 25135784
- [Background] Hasler BP, Smith LJ, Cousins JC, Bootzin RR. Circadian rhythms, sleep, and substance abuse. Sleep Med Rev. 2012 Feb;16(1):67-81. doi: 10.1016/j.smrv.2011.03.004. Epub 2011 May 26. PMID 21620743
- [Background] American Psychiatric Association (2013) Diagnostic and Statistical Manual of Mental Disorders Fifth Edition. (DSM V) 361-368.
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] HAMILTON M. A rating scale for depression. J Neurol Neurosurg Psychiatry. 1960 Feb;23(1):56-62. doi: 10.1136/jnnp.23.1.56. No abstract available. PMID 14399272
- [Background] Miller WR (1996): Form 90: A structured assessment interview for drinking and related behaviors. Center for Alcoholism: Substance Abuse and Addiction, University of New Mexico, Albuquerque.
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001 Jul;2(4):297-307. doi: 10.1016/s1389-9457(00)00065-4. PMID 11438246
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Tiffany ST, Wray JM. The clinical significance of drug craving. Ann N Y Acad Sci. 2012 Feb;1248:1-17. doi: 10.1111/j.1749-6632.2011.06298.x. Epub 2011 Dec 16. PMID 22172057
- [Background] Rush CR, Frey JM, Griffiths RR. Zaleplon and triazolam in humans: acute behavioral effects and abuse potential. Psychopharmacology (Berl). 1999 Jul;145(1):39-51. doi: 10.1007/s002130051030. PMID 10445371

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Open Label Trial of Suvorexant in Individuals With Opioid Use Disorder | Open Label Trial of Suvorexant in Individuals With Alcohol Use Disorder
Started | 6 | 22
Completed | 5 | 13
Not Completed | 1 | 9
Not completed — Withdrawal by Subject | 1 | 8
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Open Label Trial of Suvorexant in Individuals With Opioid Use Disorder | Open Label Trial of Suvorexant in Individuals With Alcohol Use Disorder | Total
Number analyzed (Participants) | 6 | 22 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.00 (10.95) | 40.91 (12.49) | 39.64 (12.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 8 | 8
  Male | 6 | 14 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 22 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 22 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Sleep Time as Measured by Actigraphy and Sleep Logs Relative to Baseline Over the Course of 7 Days of Treatment With Suvorexant in Substance Use Disorder Patients.
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Open Label Trial of Suvorexant in Individuals With Opioid Use Disorder | Open Label Trial of Suvorexant in Individuals With Alcohol Use Disorder
Number analyzed (Participants) | 4 | 14
minutes | -43.25 (61.96) | 12.68 (41.42)

2. Secondary Outcome: Relative to a Baseline, Change in Total Daily Salivary Cortisol Over the Course of 7 Days of Treatment With Suvorexant in Substance Use Disorder Patients.
Description: Saliva samples were collected at five time points each day for four days, two days at baseline (Days 1 and 2) and two days at study end (Days 7 and 8). Baseline cortisol calculated as average of Days 1 and 2; endpoint cortisol calculated as average of Days 7 and 8.
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Open Label Trial of Suvorexant in Individuals With Opioid Use Disorder | Open Label Trial of Suvorexant in Individuals With Alcohol Use Disorder
Number analyzed (Participants) | 5 | 13
ng/ml | 1.85 (9.82) | -0.58 (6.55)

3. Secondary Outcome: Relative to a Baseline, Change in Daily Reports of Craving Using Ecological Momentary Assessment (EMA Data) Over the Course of 7 Days of Treatment With Suvorexant in Substance Use Disorder Patients.
Description: The data were collected via Motorola Droid smart phones that are programmed to elicit the participants' response four times per day, during each of the 9 full study days. Change in Modified Desire for Drug Scale measured on a 100-point Likert scale (0 = no craving, 100 = maximal craving). A negative change score indicates a decrease in craving across study time.
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label Trial of Suvorexant in Individuals With Opioid Use Disorder | Open Label Trial of Suvorexant in Individuals With Alcohol Use Disorder
Number analyzed (Participants) | 5 | 11
score on a scale | -14.47 (18.43) | -8.70 (13.18)

4. Secondary Outcome: Change in Scale Items on a Modified Abuse Liability Assessment Battery Relative to Baseline.
Description: Endorsement of scale items associated with abuse liability 30 minutes after drug administration or the following morning.
  Change in Modified Abuse Liability Item Scores (0 = no change in abuse liability, 4 = maximal change in abuse liability).
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Open Label Trial of Suvorexant in Individuals With Opioid Use Disorder | Open Label Trial of Suvorexant in Individuals With Alcohol Use Disorder
Number analyzed (Participants) | 5 | 14
score on a scale
  Modified Liability Score (0-4 scale) | 0.29 (0.36) | 0.10 (0.17)
  Abuse Liability Question (use drug to get high) | 0 (0) | 0 (0)
  Abuse Liability Question (buy drug illegally) | 0 (0) | 0 (0)

ADVERSE EVENTS:
Time Frame: 10 days
Description: Subjects were routinely questioned about adverse events from nursing staff during each nightly administration.
Arm/Group | Open Label Trial of Suvorexant in Individuals With Opioid Use Disorder | Open Label Trial of Suvorexant in Individuals With Alcohol Use Disorder
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/22
Other Adverse Events (participants affected / at risk) | 3/6 | 5/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open Label Trial of Suvorexant in Individuals With Opioid Use Disorder (N=6) | Open Label Trial of Suvorexant in Individuals With Alcohol Use Disorder (N=22)
Cataplexy-like event (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label Trial of Suvorexant in Individuals With Opioid Use Disorder (N=6) | Open Label Trial of Suvorexant in Individuals With Alcohol Use Disorder (N=22)
feeling cold (General disorders) | 1 (1) | 0 (0)
tachycardia with other general disorder symptoms (General disorders) | 1 (1) | 0 (0)
vivid dreams (General disorders) | 2 (2) | 0 (0)
nightmares (General disorders) | 1 (1) | 0 (0)
inability to move (General disorders) | 1 (1) | 0 (0)
tachycardia alone (Cardiac disorders) | 1 (1) | 0 (0)
tingling in legs (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
sleepiness (General disorders) | 0 (0) | 1 (1)
headache (General disorders) | 0 (0) | 1 (1)
increased leg cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
increased elbow pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
runny nose (Infections and infestations) | 0 (0) | 1 (1)
post-nasal drip (Infections and infestations) | 0 (0) | 1 (1)
headache as part of cold (Infections and infestations) | 0 (0) | 1 (1)
feeling tired (Infections and infestations) | 0 (0) | 1 (1)
ear pain (Infections and infestations) | 0 (0) | 1 (1)
lower back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
1. Recruitment difficulties led to small numbers in the opioid use group. High number of withdrawals in the alcohol use group impacted the number of participants available for analysis.
2. For TST outcome, technical problems led to n=4 (instead of n=5) for analysis in the opioid use group. In the alcohol use group, n=13 completed the study. An additional participant completed all but one day of the study (withdrew Day 8); data was available for analysis. Total of n=14 for analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-02): https://cdn.clinicaltrials.gov/large-docs/91/NCT03412591/Prot_SAP_000.pdf
  • Informed Consent Form (2023-03-14): https://cdn.clinicaltrials.gov/large-docs/91/NCT03412591/ICF_001.pdf